CLINICAL TRIAL: NCT05230186
Title: A Tissue Collection Study in Patients Who Respond to Immune Checkpoint Inhibitors to Identify Targets of Tumor-Reactive T Cells.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-04
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor, Adult
Keywords: Solid Tumor; Renal cell carcinoma; Bladder cancer; Melanoma; Triple negative breast cancer; Colon cancer; Lung cancer; Endometrial cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Melanoma; Triple Negative Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- On-Treatment Solid Tumor Responder (Tumor Biopsy): Research tumor tissue biopsy collected at any one time point while responding to ICI therapy (radiographic regression of lesion). Tumor biopsy and companion blood sample.
  Interventions: Procedure: Tumor Biopsy
- Pre and On-Treatment Solid Tumor Responder (Tumor Biopsy): Tumor tissue collection prior to beginning ICI therapy (optional biopsy). If and when there is a response to ICI therapy, a second research tumor tissue biopsy is collected. Tumor biopsy and companion blood sample.
  Interventions: Procedure: Tumor Biopsy
- On-Treatment Solid Tumor Responder (Surgical Removal Tumor): Collection of excess tumor tissue in patients who are responding to ICI therapy and are scheduled for Surgical resection of residual disease. Excess tissue provided.
- Post-Treatment of patients with Melanoma who develop vitiligo: Up to 5 patients treated for melanoma that develop vitiligo - Skin Tissue Biopsy obtained at any point in time from any skin site with vitiligo (selected sites only). Tissue biopsy
  Interventions: Procedure: Tumor Biopsy
- On-Treatment Responder (Previously Frozen Tumor Tissue): Previously Cryopreserved Tissue obtained from a Biobank or Tissue Repository, collected from patients when they were responding to ICI Therapy (clinical data required).

INTERVENTIONS:
Procedure: Tumor Biopsy — Research biopsy of solid tumor or sharing of excess tumor tissue during a planned surgical or biopsy procedure and a companion blood sample.
  Other Names: Excess tissue during planned surgical procedure
  Groups: On-Treatment Solid Tumor Responder (Tumor Biopsy); Post-Treatment of patients with Melanoma who develop vitiligo; Pre and On-Treatment Solid Tumor Responder (Tumor Biopsy)

SUMMARY:
T Cell Receptor-engineered T-cell therapy (TCR T-cell therapy) offers a potentially transformative approach to treating cancer, but is currently limited by the lack of known targets (Maus and June, 2016; Ping et al., 2018). Arguably the most clinically meaningful way to discover new targets and TCRs for TCR T-cell therapy is to study the tumor-infiltrating lymphocytes of patients that are actively responding to immune checkpoint inhibitor (ICI) therapy. These T cells are clonally expanded as a result of checkpoint inhibition and are responsible for the patient's clinical response. The goal of this study is to acquire tumor and blood samples from up to 200 patients with solid tumor malignancies who respond to ICI therapy. T cells will be isolated from these samples and the targets of their TCRs determined using TScan's genome-wide, high-throughput target ID technology. The expected outcome of this study is the discovery of a collection of new targets for TCR T-cell therapy, along with associated TCRs that will then be developed as novel therapies for patients with similar malignancies.

ELIGIBILITY:
Inclusion Criteria:

Cohort Legend: Cohort 1: On-Treatment Responder (Biopsy), Cohort 2: Pre and On-Treatment (Biopsy), Cohort 3: On-Treatment Responder (Surgery), Cohort 4: Post-Treatment Vitiligo, Cohort 5: Post-Treatment Responder (Frozen)

1. Study Cohorts 1,2,3 and 5: Known or suspected diagnosis of non-hematological malignancy.
2. Age 18 years at time of diagnosis.
3. Research Biopsy Study Cohorts 1 and 2: ECOG performance status 0-2.
4. Ability to understand and willingness to sign an informed consent document.
5. Research Biopsy Study Cohorts 1,2,3 and 5: Patients must be eligible for or currently receiving treatment with immune checkpoint inhibitor (ICI) therapy as determined by the patient's treating oncologist. The treatment regimen may comprise more than one agent but must include at least one ICI drug. Examples of FDA-approved ICI drugs include pembrolizumab (Keytruda), nivolumab (Opdivo), atezolizumab (Tecentriq), avelumab (Bavencio), durvalumab (Imfinzi), cemiplimab (Libtayo), and ipilimumab (Yervoy). Immune-checkpoint inhibitors not on this list may also be used, provided they are FDA-approved.
6. Research Biopsy Study Cohorts 1,2,3 and 5: Patients undergoing an on-treatment biopsy must show radiographic regression of one or more lesion, as assessed by the investigator.
7. Research Biopsy Study Cohorts 1 and 2: Patients undergoing an on-treatment biopsy must have a cancer lesion that is amenable for biopsy under local anesthesia or moderate sedation per standard procedures. The tumor biopsy must have an acceptable clinical risk, as judged by the investigator.
8. Research Biopsy Study Cohorts 1,2,4: Platelet count >50,000 prior to biopsy or per the service performing the biopsy.
9. Research Biopsy Study Cohorts 1,2,4: Absolute neutrophil count >1500.
10. Research Biopsy Study Cohorts 1,2,4: Must be able to safely hold anticoagulants for 5 days prior to biopsy.
11. Research Biopsy Study Cohorts 1,2,4: Not receiving therapeutic anticoagulation at the time of the biopsy. Patients on therapeutic anticoagulation must be able to safely hold anticoagulation for the procedure with an acceptable risk, as judged by the investigator. Patients who are on anticoagulation for clinical reasons and deemed appropriate for biopsy must be OFF anticoagulation prior to biopsy as follows:

i. No warfarin (Coumadin) for 5 days. No low-molecular weight heparin (LMWH; e.g. dalteparin/ Fragmin, enoxaparin/ Lovenox) for 24 hours.

ii. No fondaparinux/ Arixtra for 48 hours. iii. Patients receiving alternative forms of anticoagulation not listed above (e.g., dabigatran, rivaroxaban, apixaban, edoxaban) should consult with the prescribing physician and the service performing the biopsy regarding safety and administration guidelines prior to biopsy. Bleeding risks with these agents should be considered when deciding on whether to perform the biopsy if for research purposes only.

Exclusion Criteria:

Cohort Legend: Cohort 1: On-Treatment Responder (Biopsy), Cohort 2: Pre and On-Treatment (Biopsy), Cohort 3: On-Treatment Responder (Surgery), Cohort 4: Post-Treatment Vitiligo, Cohort 5: Post-Treatment Responder (Frozen)

1. Concurrent disease or condition that would make the patient inappropriate for study participation, or any serious medical or psychiatric disorder that would interfere with safety.
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
3. Research Biopsy Study Cohorts 1,2,4: History of serious or life-threatening allergic reaction to local anesthetics (i.e., lidocaine, xylocaine).
4. Pregnant women are excluded because there may be an increased risk to both mother and fetus in the setting of moderate sedation, which is required for biopsies of certain anatomic sites (e.g., liver, lung, bone). Also, ionizing radiation from CT-guided biopsies may pose a risk to the unborn fetus.
5. Research Biopsy Study Cohorts 1,2,4: Active cardiac disease, defined as:

i. Uncontrolled or symptomatic angina within the past 3 months. ii. History of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes). Atrial fibrillation with controlled ventricular response on treatment is not an exclusion.

iii. Myocardial infarction < 6 months from study entry. iv. Uncontrolled or symptomatic congestive heart failure. f. Any other condition, which in the opinion of the patient's treating oncologist or the physician performing the biopsy procedure, would make participation in this protocol unreasonably hazardous for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women and members of all races and ethnic groups are eligible for this protocol. Patients with solid tumors who are responding to ICI therapy will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Single Cell Sequencing | 3 years
  Determine, through single-cell sequencing, the TCR repertoire of these tumor and blood samples to identify new targets.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Atlantic Health System, Morristown, New Jersey
  - Advanced Oncology PC, New York, New York

IPD SHARING:
Plan to Share IPD: No